CLINICAL TRIAL: NCT02337855
Title: A Phase I Study of the Safety, Reactogenicity, and Immunogenicity of Sm-TSP-2/Alhydrogel® With or Without GLA-AF for Intestinal Schistosomiasis in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 13-0009; HHSN272200800002C
Record Dates: First submitted 2015-01-08; First posted 2015-01-14 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2016-12-07

CONDITIONS: Schistosomiasis
Keywords: Intestinal; Pichia pastoris; S. mansoni; Schistosomiasis; Sm-TSP-2/Alhydrogel; Sm-TSP-2/Alhydrogel/GLA-AF; vaccine
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Group A (Experimental): N=10 subjects will receive single dose intramuscular (IM) 10mcg Sm-TSP-2/Alhydrogel® on Day1, 57 and 113
  Interventions: Biological: Sm-TSP-2/Alhydrogel
- Group B (Experimental): N=10 subjects will receive single dose intramuscular (IM) 10mcg Sm-TSP-2/Alhydrogel®/GLA-AF on Day 1, 57 and 113
  Interventions: Biological: Sm-TSP-2/Alhydrogel/GLA-AF
- Group C (Placebo Comparator): N= 4 subjects will receive single dose intramuscular (IM) Placebo (normal saline (0.9% NaCl) on Day 1, 57 and 113
  Interventions: Other: Placebo
- Group D (Experimental): N=10 subjects will receive single dose intramuscular (IM) 30mcg Sm-TSP-2/Alhydrogel® on Day 1, 57 and 113
  Interventions: Biological: Sm-TSP-2/Alhydrogel
- Group E (Experimental): N=10 subjects will receive single dose intramuscular (IM) 30mcg Sm-TSP-2/Alhydrogel®/GLA-AF on Day 1, 57 and 113
  Interventions: Biological: Sm-TSP-2/Alhydrogel/GLA-AF
- Group F (Placebo Comparator): N= 4 subjects will receive single dose intramuscular (IM) Placebo (normal saline (0.9% NaCl) on Day 1, 57 and 113
  Interventions: Other: Placebo
- Group G (Experimental): N=10 subjects will receive single dose intramuscular (IM) 100mcg Sm-TSP-2/Alhydrogel® on Day 1, 57 and 113
  Interventions: Biological: Sm-TSP-2/Alhydrogel
- Group H (Experimental): N=10 subjects will receive single dose intramuscular (IM) 100mcg Sm-TSP-2/Alhydrogel®/GLA-AF on Day 1, 57 and 113
  Interventions: Biological: Sm-TSP-2/Alhydrogel/GLA-AF
- Group I (Placebo Comparator): N= 4 subjects will receive single dose intramuscular (IM) Placebo (normal saline (0.9% NaCl) on Day 1, 57 and 113
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo: normal saline for parenteral administration. Group C. Group F, and Group I: single dose intramuscular (IM) Placebo (normal saline (0.9% NaCl) on Day 1, 57 and 113.
  Arms: Group C; Group F; Group I
Biological: Sm-TSP-2/Alhydrogel — Sm-TSP-2/Alhydrogel. Group A: single dose IM 10mcg Sm-TSP-2/Alhydrogel® on Day1, 57 and 113. Group D: single dose intramuscular (IM) 30mcg Sm-TSP-2/Alhydrogel® on Day 1, 57 and 113. Group G: single dose intramuscular (IM) 100mcg Sm-TSP-2/Alhydrogel® on Day 1, 57 and 113.
  Arms: Group A; Group D; Group G
Biological: Sm-TSP-2/Alhydrogel/GLA-AF — Sm-TSP-2/Alhydrogel/GLA-AF. Group B: single dose intramuscular (IM) 10mcg Sm-TSP-2/Alhydrogel®/GLA-AF on Day 1, 57 and 113. Group E: single dose intramuscular (IM) 30mcg Sm-TSP-2/Alhydrogel®/GLA-AF on Day 1, 57 and 113. Group H: single dose intramuscular (IM) 100mcg Sm-TSP-2/Alhydrogel®/GLA-AF on Day 1, 57 and 113.
  Arms: Group B; Group E; Group H

SUMMARY:
This is a Phase I, first-in-human study of a vaccine against S. mansoni infection.The study will recruit 72 healthy adult males and non-pregnant females from a single clinical center to test two formulations of Sm-TSP-2 vaccine (using the Alhydrogel® only, and using Alhydrogel® plus GLA-AF), each at 3 different doses: 10ug, 30ug, and 100ug. The primary objective is to assess the safety and reactogenicity of ascending doses of Sm-TSP-2/Alhydrogel® (10ug, 30ug, or 100ug) with or without GLA-AF vaccine given as three doses administered on Days 1, 57, and 113.

DETAILED DESCRIPTION:
This is a Phase I, first-in-human study of a vaccine against S. mansoni infection.The study will recruit 72 healthy adult males and non-pregnant females from a single clinical center to test two formulations of Sm-TSP-2 vaccine (using the Alhydrogel® only, and using Alhydrogel® plus GLA-AF), each at 3 different doses: 10ug, 30ug, and 100ug. The study will use a dose-escalation cohort design, in which escalation to the next dose cohort will be determined based on evaluation of pre-defined escalation criteria requiring 7 day safety data to be examined after all subjects in the current cohort have received their first dose of vaccine. For each Cohort (1-3), an initial 5 subjects (2 Sm-TSP-2/Alhydrogel®, 2 Sm-TSP-2/Alhydrogel®/GLA-AF, and 1 placebo) will be enrolled, randomized, vaccinated, and have completed Visit 2 (Day 3), before enrolling the rest of the cohort. As with dose-escalation decisions, evidence of significant reactogenicity will require further review prior to proceeding.Recruitment and enrollment into the study will occur on an ongoing basis, with each cohort being recruited and vaccinated in sequence. All subjects will be assigned investigational vaccine or placebo by randomization, and a double-blind design will be used (i.e., neither the subject nor the investigator will be aware of the study product assigned: Sm-TSP-2/Alhydrogel®, Sm-TSP-2/Alhydrogel®/GLA-AF, or placebo). Each subject will receive 3 vaccinations at Days 1, 57, and 113, and will be followed for a total of 12 months after the third dose. The study duration will be approximately 24 months, and subject participation duration will be approximately 16 months. The primary objective is to assess the safety and reactogenicity of ascending doses of Sm-TSP-2/Alhydrogel® (10ug, 30ug, or 100ug) with or without GLA-AF vaccine given as three doses administered on Days 1, 57, and 113. The secondary objectives include: (1) to assess the IgG antibody response using an indirect enzyme-linked immunosorbent assay (ELISA) at Day 127; (2) to assess the IgG antibody response using an indirect enzyme-linked immunosorbent assay (ELISA) at 14 days after dose one and two and Day 203 and 293 (3 and 6 months after the third dose) of Sm-TSP-2/Alhydrogel® (10ug, 30ug, or 100ug) with or without GLA-AF; (3) To assess the duration of the IgG antibody response using an indirect enzyme-linked immunosorbent assay (ELISA) following receipt of three doses of Sm-TSP-2/Alhydrogel® (10ug, 30ug, or 100ug) with or without GLA-AF.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria in order to be eligible for participation in this study. 1. Provide written informed consent prior to any study procedures. 2. Able to understand and comply with planned study procedures and be available for all study visits. 3. Male or non-pregnant female aged 18 to 50, inclusive. 4. Are in good health, as determined by vital signs (oral temperature, pulse, and blood pressure), medical history, and targeted physical examination based on medical history.1 Existing medical diagnoses or conditions (except those in the Subject Exclusion Criteria) must be deemed as stable chronic medical conditions. A stable chronic medical condition is defined as no change in prescription medication, dose, or frequency of medication in the last 3 months (90 days) and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months (180 days). Any change due to change of health care provider, insurance company, or that is done for financial reasons, as long as in the same class of medication, will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a violation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity. Topical, nasal, and inhaled medications (with the exception of steroids as outlined in the Subjects Exclusion Criteria), vitamins, and contraceptives are permitted. 5. Vital signs (oral temperature, pulse, and blood pressure) are all within normal protocol-defined ranges. Note: The normal protocol-defined ranges for vital signs include (a) oral temperature less than 100.0°F, (b) pulse 50 to 100 bpm, inclusive, (c) systolic blood pressure 85 to 150 mmHg, inclusive, and (d) diastolic blood pressure 55 to 90 mmHg, inclusive. 6. Laboratory tests (alanine aminotransferase, creatinine, white blood cells, hemoglobin, and platelets) are all within normal protocol-defined reference ranges.33 The normal protocol-defined ranges for laboratory tests include (a) alanine aminotransferase (ALT) of 32 IU/L or less for females or 44 IU/L or less for males, (b) creatinine 1.0 mg/dL or less for females or 1.27 mg/dL or less for males, (c) white blood cells (WBC) between 3.4 x10^3/uL and 10.8 x10^3/uL, inclusive, (d) hemoglobin 11.1 g/dL or greater for females or 12.6 g/dL or greater for males, (e) platelets between 150 x10^3/uL and 379 x10^3/uL, inclusive. Laboratory test results for 2nd and 3rd vaccinations may be at Grade 1 if considered unrelated to study product. 7. Urinalysis with no greater than trace protein and negative for glucose. 8. Female subjects of childbearing potential4 must agree to practice highly effective contraception5 for a minimum of 30 days prior to study product exposure and through 30 days after last vaccination.4 Female subjects who are surgically sterile via tubal sterilization, bilateral oophorectomy or hysterectomy or who have been postmenopausal for greater than 1 year are not considered to be of childbearing potential.5 Note: Highly effective methods of contraception are defined as having low failure rates (i.e. less than 1% per year) when used consistently and correctly and may include, but are not limited to, abstinence from intercourse with a male partner, monogamous relationship with a vasectomized partner, mal e condoms or diaphragm with spermicide, intrauterine devices, and licensed hormonal methods. 9. Female subjects of childbearing potential must have a negative urine pregnancy test within 24 hours prior to study vaccination.

Exclusion Criteria:

All subjects who meet any of the following exclusion criteria at baseline will be excluded from participation in the study. 1. Has had known infection due to S. mansoni or has traveled to an endemic area for S. mansoni infection and, during that travel, was potentially exposed to S. mansoni. 2. Has a positive urine pregnancy test prior to vaccination (if female of childbearing potential), or has the intention to become pregnant within 5 months after enrollment in this study. 3. Female subjects who are breastfeeding or plan to breastfeed at any given time from the first study vaccination until 30 days after their last study vaccination. 4. Has an acute illness, including an oral temperature of 100.0 degree F or greater, within 72 hours prior to vaccination. 5. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, diabetes, or renal disease by history, physical examination, and/or laboratory studies. 6.6 Includes the conditions and diagnoses defined as AESI in Section 9.3.3. 6. Is immunosuppressed as a result of an underlying illness or treatment.7.7 Causes for immunosuppression may include, but are not limited to, poorly-controlled diabetes mellitus, cirrhosis, renal insufficiency, active neoplastic disease or a history of any hematologic malignancy, connective tissue disease, organ transplant. 7. Using or intends to continue using oral or parenteral steroids, high-dose inhaled steroids(> 800 microg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs. 8. Positive hepatitis B surface antigen (HBsAg) 9. Positive confirmatory test for HIV infection 10. Positive confirmatory test for hepatitis C virus (HCV) infection 11. Volunteer has had a history of alcohol or illicit drug abuse during the past 24 months. 12. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 90 days prior to study vaccination. 13. History of a severe allergic reaction or anaphylaxis to known components of the vaccine 14. Has an acute or chronic medical condition that, in the opinion of the investigator, would render participation in this study unsafe or would interfere with the evaluation of responses. Note: This includes, but is not limited to: known liver disease, renal disease, neurological disorders, visual field defects, cardiac disorders, pulmonary disorders, diabetes mellitus, and transplant recipients. 15. History of splenectomy 16. Plans to undergo surgery (elective or otherwise) from the time of enrollment through 1 month post dose 3 vaccination. 17. Is participating or plans to participate in another clinical trial with an interventional agent9 during the duration of the study. Note: This may include other licensed or unlicensed vaccines, drugs, biologics, devices, blood products, or medications. 18.Received any licensed live vaccine within 30 days or any licensed inactivated vaccine within 14 days prior to the first study vaccination. Note: During influenza season, subjects will be offered seasonal influenza vaccine prior to enrollment into the study. 19. Planned receipt of any vaccine from the first study vaccination through 1 month after the last study vaccination. 20. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations. 21. Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

PRIMARY OUTCOMES:
The occurrence of new-onset chronic medical conditions (including AESI) through 12 months after the third study vaccination. | Through 12 months after the third study vaccination ( Day 478)
The occurrence of solicited injection site reactogenicity on the day of each study vaccination through 7 days after each study vaccination | Day 113-120
The occurrence of solicited injection site reactogenicity on the day of each study vaccination through 7 days after each study vaccination | Day 57-64
The occurrence of solicited injection site reactogenicity on the day of each study vaccination through 7 days after each study vaccination. | Day 1-8
The occurrence of solicited systemic reactogenicity on the day of each study vaccination through 7 days after each study vaccination. | Day 113-120
The occurrence of solicited systemic reactogenicity on the day of each study vaccination through 7 days after each study vaccination | Day 1-8
The occurrence of solicited systemic reactogenicity on the day of each study vaccination through 7 days after each study vaccination. | Day 57-64
The occurrence of study vaccine-related SAEs from the time of the first study vaccination through approximately 12 months after the last study vaccination | Day 1-12 months after the last study vaccination
The occurrence of vaccine-related clinical safety laboratory adverse events | Day 1-478

SECONDARY OUTCOMES:
The IgG antibody response using an indirect enzyme-linked immunosorbent assay (ELISA) on the day of each dose, 14 days after each dose, and 3 and 6 months after the third dose of Sm-TSP-2/Alhydrogel (10ug, 30ug, or 100ug) with or without GLA-AF | Days 1, 5, 57, 71, 113,127, 203 and 293
The IgG level using an indirect enzyme-linked immunosorbent assay (ELISA) at Day 127 | Day 127

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas, United States